CLINICAL TRIAL: NCT04743869
Title: Calcium Phosphate Versus PMMA Cement in Unstable Thoracolumbar Burst Fractures Treated With Dorsal Instrumentation in Patients > 50 Years of Age Randomized Controlled Non-inferiority Trial Design
Brief Title: Calcium Phosphate Versus PMMA Cement in Thoracolumbar Fractures
Acronym: CaPvsPMMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V 2.0
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: SPINAL Fracture
Keywords: Spinal Fractures; Fractures; Polymethyl Methacrylate; PMMA; Bone Cements; Calciumphosphate; Thoracolumbar Fractures; Dorsal Instrumentation; Burst Fractures; Balloon Kyphoplasty
MeSH Terms: conditions — Spinal Fractures; Fractures, Bone

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients and study nurse will be blinded to treatment allocation; however, surgeons cannot be blinded due to different techniques of bone cement application. A centralized and automated internet-based randomization system will ensure concealed randomization of study participants. Participants will be the unit of randomization. Randomization will be carried out with randomizer.at and will occur prior to the surgical procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KYPHON® ActivOs™10 Bone Cement with hydroxyapatite (Active Comparator): As a reference device KYPHON® ActivOs™10 Bone Cement with hydroxyapatite (Medtronic) for treatment of vertebral compression fractures will be used. It is a polymethylmethacrylate (PMMA) bone cement containing hydroxyapatite (HA) for use in the treatment of patients with vertebral compression fractures (VCFs) who are undergoing minimally invasive surgery with KYPHON® Balloon Kyphoplasty. This bone substitute has already been approved and is in use in the patients at the age of 50 or older.
  Interventions: Device: KYPHON ActivOs® Bone Cement with Hydroxyapatite
- KyphOs FS™ (Experimental): The test device KyphOs FS™ will be used in patients at the age of 50 and older in order to prove its superiority over the currently used PMMA bone cement.
  Interventions: Device: Kyphos FS™ Bone Substitute

INTERVENTIONS:
Device: Kyphos FS™ Bone Substitute — Dorsal instrumentation via Longitude II (Medtronic Austria GmbH/Vienna) and balloon kyphoplasty are performed. KyphOs FS™ bone cement will be introduced in the fractured vertebral body.
  Other Names: KyphOs FS™ Bone Cement; KyphOs FS™ Medtronic Spine LLC, Minneapolis, MN, USA
  Arms: KyphOs FS™
Device: KYPHON ActivOs® Bone Cement with Hydroxyapatite — Dorsal instrumentation via Longitude II (Medtronic Austria GmbH/Vienna) and balloon kyphoplasty are performed. KYPHON ActivOs® Bone Cement with Hydroxyapatite will be introduced in the fractured vertebral body.
  Other Names: KYPHON ActivOs® Bone Cement with Hydroxyapatite, Medtronic Spine LLC, Minneapolis, MN, USA
  Arms: KYPHON® ActivOs™10 Bone Cement with hydroxyapatite

SUMMARY:
Patients at the age of 50 or older presenting with thoracolumbar fractures including segments TH 6-L5 and A3/A4 fractures according to the AO Spine fracture classification after the acute trauma and planned surgery within 3 weeks following trauma will be asked to participate in a randomized trial in which they will receive either Calciumphosphate (CaP) or Polymethylmethacrylate (PMMA) as part of a standardized treatment approach. Regardless of the group patients are randomized to, all participating patients undergo the same surgical procedure except for the preparation and administration of bone cement. The study participation period for each patient is 1 year from the date of the surgery and includes 4 defined time points that include follow-up clinical visits for imaging and progress checks at 6 weeks, 3 months, 6 months and 12 months after surgery. At each follow-up visit, a combination of questionnaires and radiological imaging will be performed to assess general health status, disability level and pain control, as well as objective results of the surgery. The main outcome measure will be the loss of correction rate that will be measured through the bi-segmental COBB angle presented in the CT-scan.

ELIGIBILITY:
Inclusion Criteria:

* Written consent of the participant after being informed
* Acute trauma (surgery within three weeks following trauma)
* Thoracolumbar fractures including segments TH 6-L5
* A3/A4 fractures according to the AO Spine fracture classification
* Patient age ≥ 50 years
* Minimum follow up 1 year

Exclusion Criteria:

* Presence of neurological deficits at the time of surgery
* Pathological fractures (bone metastases)
* Traumatic brain injury
* Ankylosing spondylitis as a comorbidity
* Pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
The change in correction rates when using CaP | Preoperatively (determination of fracture classification), postoperatively (immediately following surgery), 1 year postoperatively
  The main outcome measure 1 will be the loss of correction rate that will be measured through the bi-segmental COBB angle presented in the CT-scan. The Cobb angle will be measured between the superior end plate of the vertebral body cephalad to the injury and the inferior end plate of the vertebral body caudal to the injury.
The change in correction rates when using PMMA | Preoperatively (determination of fracture classification), postoperatively (immediately following surgery), 1 year postoperatively
  The main outcome 2 measure will be the loss of correction rate that will be measured through the bi-segmental COBB angle presented in the CT-scan. The Cobb angle will be measured between the superior end plate of the vertebral body cephalad to the injury and the inferior end plate of the vertebral body caudal to the injury. Measurements will be taken from CT scans.

SECONDARY OUTCOMES:
The change in vertebral body height when using CaP | Preoperatively, postoperatively (immediately following the surgery), 1 year postoperatively
  The percentage loss of the vertebral body height will be calculated by dividing the height of the fractured vertebra by the average height of the cephalad and caudad vertebrae and then subtracting this number from 100%. Measurements will be taken from CT scans.
The change in vertebral body height when using PMMA | Preoperatively, postoperatively (immediately following the surgery), 1 year postoperatively
  The percentage loss of the vertebral body height will be calculated by dividing the height of the fractured vertebra by the average height of the cephalad and caudad vertebrae and then subtracting this number from 100%.
Changes in complication rates when using PMMA | 6 weeks, 3 months, 6 months and 12 months postoperatively
  The occurence of the complication rates, in particular cement extravasation and temporary fall in blood pressure, will be compared between the two groups for each time point using the Student´s t-test for independent samples. In addition, a paired Student´s t-test will be performed within each group in order to evaluate the differences in means of the secondary endpoints measured at the defined timepoints.
Changes in complication rates when using CaP | 6 weeks, 3 months, 6 months and 12 months postoperatively
  The occurence of the complication rates, in particular cement extravasation and temporary fall in blood pressure, will be compared between the two groups for each time point using the Student´s t-test for independent samples. In addition, a paired Student´s t-test will be performed within each group in order to evaluate the differences in means of the secondary endpoints measured at the defined timepoints.
Change in the disability on the ODI rating scale in patients with PMMA | Five times - after the surgery, at each study visit (6 weeks, 3 months, 6 months and 12 months postoperatively)
  ODI is mainly used in spine trauma patients. A score of 0% to 20% indicates minimal disability; 21% to 40%, moderate disability; and 41% to 60% severe disability.
Change in the disability on the ODI rating scale in patients with CaP | Five times - after the surgery, at each study visit (6 weeks, 3 months, 6 months and 12 months postoperatively)
  ODI is mainly used in spine trauma patients. A score of 0% to 20% indicates minimal disability; 21% to 40%, moderate disability; and 41% to 60% severe disability.
Change in pain on the spine VAS in patients with PMMA | Five times - after the surgery, at each study visit (6 weeks, 3 months, 6 months and 12 months postoperatively)
  VAS - Spine Visual Analogue Scale is a measurement that measures pain intensity and it is completed by patients themselves.
Change in pain on the spine VAS in patients with CaP | Five times - after the surgery, at each study visit (6 weeks, 3 months, 6 months and 12 months postoperatively)
  VAS - Spine Visual Analogue Scale is a measurement that measures pain intensity and it is completed by patients themselves.
Change in quality of life in patients with PMMA measured by the 36-item Short Form Survey | Five times - after the surgery, at each study visit (6 weeks, 3 months, 6 months and 12 months postoperatively)
  The 36-Item Short Form Survey (SF-36) will be used to assess patient´s self-reported quality of life.
Change in quality of life in patients with CaP measured by the 36-item Short Form Survey | Five times - after the surgery, at each study visit (6 weeks, 3 months, 6 months and 12 months postoperatively)
  The 36-Item Short Form Survey (SF-36) will be used to assess patient´s self-reported quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Puchwein, Assist.Prof., Principal Investigator — University Hospital Graz

IPD SHARING:
Plan to Share IPD: No
Results of the study are planned to be made public within a scientific work.